CLINICAL TRIAL: NCT07350057
Title: Phase Ib Study on the Prevention of Graft-versus-host Disease (GVHD) in Children After Haploid Stem Cell Transplantation Using Cyclophosphamide (PTCy) Combined With Sirolimus and VIC-1911 Tablets
Brief Title: A Preliminary Clinical Study on the Efficacy of Cyclophosphamide and Sirolimus Combined With VIC-1911 in Preventing Graft-versus-Host Disease After Haploidentical Stem Cell Transplantation in Children
Acronym: GVHD
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, wang xiaodong, Principal Investigator, Shanghai Children's Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: JSI-1911-103
Record Dates: First submitted 2025-12-19; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-07

CONDITIONS: GVHD (Acute or Chronic)
MeSH Terms: conditions — Graft vs Host Disease; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Phase Ib Study of Post-Transplant Cyclophosphamide (PTCy) Combined with Sirolimus and VIC-1911 Table (Experimental)
  Interventions: Drug: 1mg /kg VIC-1911

INTERVENTIONS:
Drug: 1mg /kg VIC-1911 — VIC-1911 D5-D45 1mg/kg（maximum 75mg）Oral administration on an empty stomach Bid VIC-1911 D5-D45 1.25mg/kg（maximum 75mg）Oral administration on an empty stomach Bid VIC-1911 D5-D45 0.75mg/kg（maximum 75mg）Oral administration on an empty stomach Bid
  Other Names: 1.25mg/kg VIC-1911

SUMMARY:
This study is a single arm, open label Phase Ib clinical trial, consisting of two parts: the first part is a safety introduction trial, and the second part is a dose escalation trial. In the first part, the tolerability, safety, PK characteristics, PD characteristics, and preliminary efficacy of VIC-1911 tablets in combination with PTCy and sirolimus will be explored. The first part will conduct safety introduction tests at the same dose as those already tested abroad to determine the dosage required for VIC-1911 tablets to meet safety and effective biological activity. The dose limiting toxicity (DLT) in Phase I study will be evaluated from the first administration of VIC-1911 tablets to 28 days after administration. On this basis, the second part of the experiment will be conducted to further explore the effectiveness and safety of VIC-1911 tablets combined with PTCy and sirolimus under RP2D for preventing GVHD in haplo HSCT patients after myeloablative pretreatment

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all of the following criteria in order to participate in this study:

  1. Children aged 8-18, regardless of gender;
  2. Prior to the start of the study, the subjects and their legal guardians shall sign a written informed consent form;
  3. Patients diagnosed with the following blood diseases and deciding to undergo haplo HSCT:

     1. Patients diagnosed with acute myeloid leukemia or high-risk acute lymphoblastic leukemia who have achieved complete remission (CR) through induction therapy;;
     2. Patients diagnosed with myelodysplastic syndrome (MDS) and with an International Prognostic Scoring System (IPSS, please refer to Appendix 1a) score of medium risk 2 or high risk, or with severe blood cell reduction in the IPSS low-risk group, who have undergone ineffective treatment or have poor prognosis due to genetic abnormalities (such as -7,3q26 rearrangement, TP53 gene mutation, complex karyotype, monomeric karyotype);
  4. There are peripheral blood stem cell donors who are 5/10 HLA haploidentical;
  5. Karnofsky (KPS) score (see Appendix 2) ≥ 80 points;
  6. Possess sufficient organ functions, including:

     1. Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or calculated creatinine clearance rate (using Cockcroft Gault formula, please refer to Appendix 3) ≥ 50ml/min;
     2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) are both ≤ 2 × ULN, and total bilirubin is<1.5 × ULN (for subjects with Gilbert syndrome, inclusion should be determined by researchers and medical monitors);
     3. Ferritin<2000ng/ml;
     4. Adequate lung function, defined as FEV1, FVC, DLCO ≥ 50% of expected values; Pulmonary function test: FEV1, FVC, DLCO ≥ 50% of expected values;
     5. Adequate cardiac function, defined as a left ventricular ejection fraction (LVEF) of ≥ 45% evaluated through echocardiography or multiple uptake gated acquisition (MUGA) scans;

Exclusion Criteria:

* Subjects who meet any of the following criteria will be excluded from participating in this study:

  1. Hematopoietic stem cell transplantation comorbidity index (HCT-CI)>4 (Sorror criteria, please refer to Appendix 5);
  2. Plan to start post transplant maintenance treatment within 75 days after transplantation;
  3. Those who are allergic to cyclophosphamide, VIC-1911 tablets, sirolimus, and sirolimus derivatives, or any excipient component of the above drugs;
  4. Those who are unable or unwilling to discontinue other immunosuppressive treatments before the start of the study;
  5. History of eye diseases, patients with central or branch retinal artery or vein occlusion, accompanied by significant visual impairment, or other retinal diseases determined by ophthalmologists leading to visual impairment;
  6. Have a serious history of cardiovascular and cerebrovascular diseases, including but not limited to:

     1. Hypertension that cannot be controlled after standard clinical treatment (systolic blood pressure>160mmHg or diastolic blood pressure>100mmHg for more than 4 weeks);
     2. Severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, II-III degree atrioventricular block, etc; According to the standards of the New York Heart Association (NYHA) in the United States (please refer to Appendix 6), patients with III-IV grade heart failure;
     3. Within 6 months prior to the first administration, any of the following conditions have occurred: myocardial infarction, severe/unstable angina, persistent arrhythmia with CTCAE v5.0 ≥ 2, atrial fibrillation of any grade, coronary/peripheral artery bypass surgery, symptomatic congestive heart failure with CTCAE v5.0 ≥ 2, cerebrovascular accident (note: patients with lacunar cerebral infarction may be considered for inclusion);
     4. Any factors that increase the risk of QTc interval prolongation or arrhythmia, such as heart failure, hypokalemia, congenital long QT syndrome, or the use of any known concomitant medication that may prolong the QT interval (see Appendix 7), except for antibiotics used for the prevention or treatment of infections;
  7. Those who have undergone major surgical procedures within 28 days prior to administration, or those who are expected to undergo major surgery during the trial period;
  8. During screening, there are clinically significant gastrointestinal abnormalities that may affect the intake, transport, or absorption of drugs (such as swallowing difficulties, uncontrollable nausea and vomiting, active gastric ulcers, ulcerative colitis, Crohn's disease, chronic diarrhea, intestinal obstruction, etc.);
  9. Have received the drug used in clinical trials or are currently participating in clinical trials involving the drug within 28 days before administration or within 5 half lives of the drug (whichever is longer);
  10. People who have difficulty with venous blood collection;
  11. Individuals who are positive for hepatitis B surface antigen (HBsAg) and/or core antibodies and positive for hepatitis B virus deoxyribonucleic acid (HBV DNA), positive for hepatitis C virus (HCV) antibodies and positive for hepatitis C virus ribonucleotide (HCV RNA) testing, positive for Treponema pallidum antibodies, and positive for human immunodeficiency virus antibodies (HIV Ab) during screening;
  12. Subjects who have used appropriate antibiotics or other treatments but still have uncontrolled systemic fungal, bacterial, viral, or other infections;
  13. Have undergone major organ surgery (excluding aspiration biopsy) or severe trauma within 4 weeks prior to the first administration, or require elective surgery during the trial period;
  14. The researchers believe that the patient is not suitable to participate in this study (such as not meeting the most beneficial treatment for the patient, patient compliance, etc.).

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Estimated)
Dates: Start 2026-03-25 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
1.Determine the recommended phase 2 dose (RP2D) of VIC-1911 tablets combined with post transplant cyclophosphamide (PTCy) and sirolimus for the prevention of GVHD in haplo HSCT pediatric patients (Only evaluated in Part 1) | Expected 2 years
  1. The incidence of dose limiting toxicity (DLT) during observation period;
  2. When used in combination, the RP2D of VIC-1911 tablets. The dose of RP2D should achieve the minimum expected biological efficacy, and the incidence of DLT in patients at this dose should be less than 30%. The minimum expected biological efficacy is 65% of patients with CD4+pH3ser10+T cells<54% at baseline by day 21 (-3 to+7), based on the lower confidence interval of pre transplant CD4+pH3ser10+T cell frequency (note: pH3ser10 is the phosphoprotein target of Aurora kinase A)